CLINICAL TRIAL: NCT03374852
Title: A Phase II Open-Label Clinical Trial of CPI-613 in Combination With Modified FOLFIRINOX in Patients With Locally Advanced Pancreatic Cancer and Good Performance Status
Brief Title: CPI-613 in Combination With Modified FOLFIRINOX in Patients With Locally Advanced Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Left institution on 8/6/2018 and study has been final reported with IRB. Never opened to accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18P.087; JT 11772 (Other: JeffTrial Number)
Record Dates: First submitted 2017-12-04; First posted 2017-12-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-613 + mFOLFIRNOX (Experimental): CPI-613: 500 mg/m2, IV infusion at a rate of 4 mL/min via a central venous port mFOLFIRNOX (given immediately after CPI-613 administration): Oxaliplatin (Eloxatin) at 65 mg/m2 given as a 2-hr IV infusion via a central venous port
  * Folinic acid at 400 mg/m2 given as a 90-min infusion immediately after oxaliplatin, and concurrently with irinotecan (Camptosar).
  * Irniotecan at 140 mg/m2 given as a 90-min IV infusion via a central venous port via a Yconnector.
  * Flurouracil (5FU) at 400 mg/m2 as bolus followed by a 46-hr infusion at 2400 mg/m2, starting immediately after completion of folinic acid and irinotecan
  Interventions: Drug: CPI-613; Drug: mFOLFIRNOX

INTERVENTIONS:
Drug: CPI-613 — 500 mg/m2, IV infusion at a rate of 4 mL/min via a central venous port
Drug: mFOLFIRNOX — mFOLFIRNOX (given immediately after CPI-613 administration):

SUMMARY:
This study is a single arm, phase II trial, of 45 patients with locally advanced pancreatic ductal adenocarcinoma. The efficacy of the novel drug and mitochondrial inhibitor, CPI-613, in conjunction with standard-of-care FOLFRINOX, as a first-line therapy will be evaluated. Pre-treatment, diagnostic biopsy tissue will be collected when available, and clinical data will be evaluated to determine if the combination results in improved overall survival compared to historical experience.

DETAILED DESCRIPTION:
Primary Objective:

1) To determine if CPI-613 increases overall survival (OS) when used in combination with mFOLFIRINOX, in patients with locally advanced pancreatic cancer.

Secondary (Exploratory) Objectives:

1. To assess the safety of CPI-613 + mFOLFIRINOX combination in patients with locally advanced pancreatic cancer.
2. To collect tissue specimens for future correlative studies
3. To estimate median progression free survival (PFS) when CPI- 613 is used in combination with mFOLFIRINOX, in patients with locally advanced pancreatic cancer.
4. To estimate the percent resected when CPI-613 is used in combination with mFOLFIRINOX in patients with locally advanced pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Cytologically confirmed pancreatic adenocarcinoma
* Locally advanced (including unresectable or borderline resectable) pancreatic cancer based on CT imaging, as determined by the PI
* Eastern Cooperative Oncology Group (ECOG) performance status being 0-1 within 1 week of planned start of therapy.
* Expected survival >3 months.
* Male and female patients 18 to not older than 80 years of age
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device (IUD), oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
* Laboratory values ≤2 weeks must be:

  * Adequate hematologic (granulocyte count ≥1500/mm3; white blood cell [WBC] ≥3500 cells/mm3; platelet count ≥100,000 cells/mm3; absolute neutrophil count [ANC] ≥1500 cells/mm3; and hemoglobin ≥9 g/dL).
  * Adequate hepatic function (aspartate aminotransferase [AST/SGOT] ≤3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] ≤3x UNL, bilirubin ≤1.5x UNL).
  * Adequate renal function (serum creatinine ≤2.0 mg/dL or 177 μmol/L).
  * Adequate coagulation ("International Normalized Ratio" or INR must be <1.5) unless on therapeutic blood thinners.
* No evidence of clinically significant active infection and no serious infection within the past month.
* Mentally competent, ability to understand and willingness to sign the informed consent form.

Exclusion Criteria:

* Patients under the age of 18 or older than 80 years of age
* Endocrine or acinar pancreatic carcinoma
* Resectable pancreatic cancer
* Metastatic pancreatic cancer based on imaging
* Prior surgical or medical treatment for pancreatic cancer
* Patients receiving any other standard or investigational treatment for their cancer with a primary goal of improving survival within the past 2 weeks prior to initiation of CPI-613 treatment.
* Serious medical illness that would potentially increase patients' risk for toxicity
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease).
* Pregnant women, or women of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown).
* Lactating females.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Life expectancy less than 3 months.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.
* Unwilling or unable to follow protocol requirements.
* Active including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, or symptomatic myocardial infarction.
* Patients with a history of myocardial infarction that is <3 months prior to registration.
* Evidence of active infection, or serious infection within the past month.
* Patients with known HIV infection.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-10-05 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Enrollment to death
  Overall survival defined as the interval between enrollment and death.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression free survival time is defined as time from enrollment until progression or death. The distribution of PFS will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Winter, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/